CLINICAL TRIAL: NCT01980810
Title: Pase 2 Study of Albumin-bounded Paclitaxel Plus S-1 as First-line Chemotherapy for Locally Advanced or Metastatic Gastric or Gastro-esophageal Adenocarcinoma
Brief Title: First Line Chemotherapy for Advanced Cancer
Acronym: GC-A-003
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruit too slowly
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Lin Yang, professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-037-nab
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Albumin-Bound Paclitaxel; Taxes; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- albumin-bounded paclitaxel plus S-1 (Experimental): arm 1:albumin-bounded paclitaxel 200mg iv d1 and S-1 80mg/m2/d po d1-10, repeated every 2 weeks,up to 9 cycles,then S-1 as single agent to treat to disease progression
  Interventions: Drug: albumin-bounded paclitaxel; Drug: S-1

INTERVENTIONS:
Drug: albumin-bounded paclitaxel — 200mg iv d1, repeat every 2 weeks,until disease progression,or up to 9 cycles
  Other Names: Abraxane; Paclitaxel Albumin-stabilized Nanoparticle Formulation
Drug: S-1 — 40mg/m2 po, bid,d1-10,repeated every 2 weeks until disease progression
  Other Names: TS-1

SUMMARY:
The purpose of this study is to determine whether albumine-bounded paclitaxel plus S-1 are effective in the treatment of advanced gastric or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
This phase II study was designed to evaluate the efficacy and safety of albumin-bounded paclitaxel combined with S-1 as first-line chemotherapy for inoperable and /or metastatic gastric or gastroesophageal junction cancer.Primary endpoint was overall response rate.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable locally advanced, recurrent, and/or metastatic adenocarcinoma of the stomach or gastro-esophageal junction
* Adult patients >=18 years of age
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-2;
* At least have one measurable disease(according to RECIST)
* Adequate bone marrow,renal and liver function

Exclusion Criteria:

* Previous chemotherapy for advanced/metastatic disease
* Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-09; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
response rate | 12 weeks

SECONDARY OUTCOMES:
progression free survival | 1 year
overall survival | 1 year
number of adverse event | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, MD, Principal Investigator — Department of medical oncology,Cancer hospital and institute,CAMS
Locations (1):
- Department of Medical Oncology,Cancer Hostpital and Institute,CAMS, Beijing, China